CLINICAL TRIAL: NCT01348672
Title: Prospective Study Phase: Retinal Oxygen Saturation, Blood Flow, Vascular Function and High Resolution Morphometric Imaging in the Living Human Eye
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Toronto (Other)
Collaborators: Ontario Research Fund (Other)
Responsible Party: Principal Investigator, Chris Hudson, Professor, University of Toronto
Other Study IDs: ORF2
Record Dates: First submitted 2011-02-27; First posted 2011-05-05 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Age Related Macular Degeneration; Glaucoma; Diabetic Retinopathy.
Keywords: Age related macular degeneration; Glaucoma; Diabetic retinopathy; Retinal oxygen saturation; Blood flow; Vascular function; High resolution imaging
MeSH Terms: conditions — Macular Degeneration; Glaucoma; Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1. ARMD Study arm: The ARMD study arm (n=150) consists of 3 groups. The groups are organised according to established risk criteria for clinical progression (AREDS, 2003).
  Group 1A (n=50); Early stage ARMD with low risk of progression; several small drusen, or a few medium-sized drusen, in one or both eyes. One eye will be randomly selected for the study.
  Group 2A (n=50); Intermediate ARMD with high risk of progression to advanced ARMD; many medium-sized drusen, or one or more large drusen, in one or both eyes. More severely affected eyewill be selected for the study.
  Group 3A (n=50); In one eye only, either a break-down of light-sensitive cells and supporting tissue in the central retinal area (i.e. geographic atrophy), or abnormal and fragile blood vessels under the retina (i.e. choroidal neovascular membrane formation). The fellow eye is at high risk of progression to advanced ARMD. The fellow eye will be selected for the study.
- 2. POAG study arm: Patient groups are organised according to established risk criteria for clinical progression (EMGT, 2003).
  Group 1P (n=36); Stable, early to moderate, treated patients with POAG. Early to moderate POAG is defined as having an untreated IOP prior to treatment of >21mmHg and a repeatable visual field defect with a Mean Deviation of <12dB and/or documented but stable ONH appearance, consistent with a diagnosis of glaucoma.
  Group 2P (n=36); Early to moderate, treated patients with normal tension glaucoma (NTG). Normal Tension Glaucoma is defined using the same criteria as POAG but with an untreated IOP of <21mmHg throughout the day. This group has NTG and is thought to be at increased risk of vascular dysfunction due to loss of ONH perfusion.
  Group 3P (n=36); Early to moderate, treated patients with POAG or NTG with recurrent disc hemorrhage (indicative of progression).
- 3. DR study arm: DR patient groups are organised according to established risk factors for the clinical progression of DR (increasing from Groups 1 A to 3 A, ETDRS, 1991). We will recruit 41 patients per group (Klein et al, 1984).
  Group 1D (n=41); Type 2 diabetic patients with no, or minimal, clinically visible DR. These patients are at low risk of developing sight-threatening DR.
  Group 2D (n=41); Type 2 diabetic patients with microaneurysms and / or hard exudates within 2 disc diameters of the fovea and no clinical evidence of retinal thickening. These patients are at increased risk of developing DME.
  Group 3D (n=41); Type 2 diabetic patients with the typical features of moderate-to-severe DR i.e. venous beading, intra-retinal microvascular abnormalities (IRMA) and dark blot intra-retinal haemorrhages. These patients are at a much increased risk of developing proliferative DR and/or ischemic maculopathy.

SUMMARY:
Canadians fear loss of vision more than any other disability. Vision loss has an enormous impact on quality-of-life and is extremely costly from a societal and economic perspective. In 2001, more than 600,000 Canadians were estimated to have severe vision loss, accounting for 17% of total disability in Canada. One in 9 individuals experience severe vision loss by 65 years of age; however, this increases to 1 in 4 individuals by 75 years. The financial cost of vision loss in Canada is $15.8 billion per year. There is a general perception that vision loss is "normal with aging" but 75% of vision loss is estimated to be preventable. The major causes of severe vision loss are age-related macular degeneration (ARMD), glaucoma, particularly primary open-angle glaucoma (POAG), and diabetic retinopathy (DR). Canada is headed for an epidemic of age-related eye disease and, unless something is done to prepare for this, severe vision loss will have significant consequences in terms of societal and economic costs. Through this proposed Research Program, and in conjunction with the investigators international academic and private sector partners, the investigators will build and develop unique quantitative imaging technologies to permit non-invasive assessment of visual changes, structural changes in the thickness of the retina at the back of the eye and also changes in the amount of blood flowing through the blood vessels that feed the retina with oxygen. This research will add to the investigators basic knowledge in predicting the development of sight-threatening change in patients with the three diseases, and facilitate earlier detection of the problem to help us discover earlier treatments for people with these conditions. The reliability of each imaging technology will be assessed by determining its ability to differentiate between diseased and healthy eyes. Cross-sectional analyses at yearly intervals, as well as change over time analyses, will be undertaken.

DETAILED DESCRIPTION:
This research will add to our basic knowledge in predicting the development of sight-threatening change in patient with the ARMD, diabetic retinopathy and primary open glaucoma, and facilitate earlier detection of the problem to help us discover earlier treatments for people with these conditions. The reliability of each imaging technology will be assessed by determining its ability to differentiate between diseased and healthy eyes. Through this proposed Research Program, and in conjunction with our international academic and private sector partners, we will build and develop unique quantitative imaging technologies to:

* Comprehensively assess the blood supply to, and vascular regulation characteristics of the posterior segment of the eye, a diagnostic capability that is currently severely limited.
* Assess oxygen saturation disturbances in the retina and ON that occur prior to clinically detectable changes, diagnostic capability that currently does not exist
* Using the retinal blood supply and oxygen saturation parameters, we will derive net oxygen delivery to the retina and optic nerve head (ONH), a diagnostic capability that does not exist.

ELIGIBILITY:
Inclusion criteria:

* Subjects diagnosed with age related macular degeneration
* Subjects diagnosed with glaucoma
* Subjects diagnosed with diabetic retinopathy

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The cohorts will be selected from the clinics of retinal and glaucoma specialists at the Toronto Western Hospital and will be identified from their charts. Clinicians will ask eligible patients whether they would be interested in participating.
  Also flyers advertising the study will be posted at Toronto Western Hospital and anyone interested can contact the principal investigator.
Sampling Method: Non-Probability Sample
Enrollment: 381 (Estimated)
Dates: Start 2012-03; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Cross-sectional relationship between retinal / ON oxygen saturation, vascular dysregulation and retinal morphometry | 5 years
  To investigate the cross-sectional relationship between retinal / ON oxygen saturation, vascular dysregulation and retinal morphometry in groups of patients at risk of progres
Prospective relationship between retinal/ON oxygen saturation disturbances, vascular dysregulation, retinal morphometry and clinical outcomes | 5 years
  To establish the prospective relationship between retinal/ON oxygen saturation disturbances, vascular dysregulation, retinal morphometry and clinical outcomes in patients at risk of progression of ARMD, POAG and DR and age-matched healthy controls
Topographic distribution of retinal / ON oxygen saturation disturbance, vascular dysfunction and change in morphometric parameters | 5 years
  To investigate the topographic distribution of retinal / ON oxygen saturation disturbance, vascular dysfunction and change in morphometric parameters in groups of patients at risk of progression of ARMD, POAG and DR

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Hudson, OD, PhD, Principal Investigator — Toronto Western Hospital, Toronto Western Research Institute, University of Toronto, University of Waterloo
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Bressler NM, Bressler SB, Congdon NG, Ferris FL 3rd, Friedman DS, Klein R, Lindblad AS, Milton RC, Seddon JM; Age-Related Eye Disease Study Research Group. Potential public health impact of Age-Related Eye Disease Study results: AREDS report no. 11. Arch Ophthalmol. 2003 Nov;121(11):1621-4. doi: 10.1001/archopht.121.11.1621. PMID 14609922
- [Background] Klein R, Wang Q, Klein BE, Moss SE, Meuer SM. The relationship of age-related maculopathy, cataract, and glaucoma to visual acuity. Invest Ophthalmol Vis Sci. 1995 Jan;36(1):182-91. PMID 7822146
- [Background] Fundus photographic risk factors for progression of diabetic retinopathy. ETDRS report number 12. Early Treatment Diabetic Retinopathy Study Research Group. Ophthalmology. 1991 May;98(5 Suppl):823-33. PMID 2062515
- [Background] Klein R, Klein BE, Moss SE, Davis MD, DeMets DL. The Wisconsin epidemiologic study of diabetic retinopathy. III. Prevalence and risk of diabetic retinopathy when age at diagnosis is 30 or more years. Arch Ophthalmol. 1984 Apr;102(4):527-32. doi: 10.1001/archopht.1984.01040030405011. PMID 6367725
- [Background] Leske MC, Heijl A, Hussein M, Bengtsson B, Hyman L, Komaroff E; Early Manifest Glaucoma Trial Group. Factors for glaucoma progression and the effect of treatment: the early manifest glaucoma trial. Arch Ophthalmol. 2003 Jan;121(1):48-56. doi: 10.1001/archopht.121.1.48. PMID 12523884